CLINICAL TRIAL: NCT01045980
Title: The Effect of Bio-impedance Analysis and Vitamin D Versus Usual Care on Left Ventricular Mass in Peritoneal Dialysis Patients: a Randomized Controlled Trial
Brief Title: Assessment of Bioimpedance and Vitamin D and LV Mass in PD Patients (FLUID Study)
Acronym: FLUID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SJH-Renal-RCT-003
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Disorders Associated With Peritoneal Dialysis
Keywords: Peritoneal dialysis; Impedance, bioelectric; Hypertrophy, left ventricular; Fluid status; Volume overload; Congestive heart failure; Cardiovascular outcomes; Randomized controlled trial
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Edema; Heart Failure | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bioimpedance and Vitamin D (Experimental): Bioimpedance and Vitamin D
  Interventions: Drug: Bioimpedance and Vitamin D
- Usual care and Vitamin D (Experimental): Usual Care and Vitamin D3
  Interventions: Drug: Usual care and Vitamin D
- Bioimpedance and Placebo (Experimental): Bioimpedance and Placebo
  Interventions: Device: Bioimpedance and Placebo
- Usual Care and Placebo (Placebo Comparator): Usual Care and Placebo
  Interventions: Drug: Usual care and placebo

INTERVENTIONS:
Drug: Bioimpedance and Vitamin D — Intervention subjects will undergo BIA assessment monthly for 1 year, and then every 3 months until the end of the planned 3-year study. Protocolized interventions to achieve euvolemia will occur based on the BIA result and they include sodium restriction, addition of diuretics, use of icodextrin, and additional rational changes to the PD prescription.
  Arms: Bioimpedance and Vitamin D
Drug: Usual care and placebo — Usual care (not bioimpedance guided volume management) and Placebo
  Arms: Usual Care and Placebo
Drug: Usual care and Vitamin D — Usual care (not bioimpedance guided volume management) and Vitamin D
  Arms: Usual care and Vitamin D
Device: Bioimpedance and Placebo — Bioimpedance guided volume management and Placebo
  Arms: Bioimpedance and Placebo

SUMMARY:
The main purpose of this study is to compare the effects of using bio-impedance analysis to guide management of fluid status versus routine clinical care on heart structure. In addition, Vitamin D is being assessed to determine its effect on heart structure.

DETAILED DESCRIPTION:
Patients on peritoneal dialysis are frequently hypervolemic which is associated with deleterious changes in left ventricular (LV) architecture including increased LV mass. In dialysis patients, increased LV mass is associated with death. Recent randomized trials have demonstrated that increasing small solute clearance is not associated with improved outcomes - hence an increased interest in the management of volume control in ESRD patients. Bioimpedance analysis is inexpensive, safe and easy to use and appears to be more useful than other techniques to assess volume status in dialysis patients. In addition, dialysis patients are vitamin D deficient and this is also associated with an increased LV mass and its inherent complications.

This study will evaluate the use of bioimpedance analysis versus usual care to assess and manage volume status and the use of vitamin D versus placebo in peritoneal dialysis patients and its effect on LV mass as measured by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* on peritoneal dialysis

Exclusion Criteria:

* Contraindication to MRI including presence of a pacemaker, defibrillator, ferromagnetic cerebral aneurysm clips, cochlear implants or eye prosthesis, neurostimulators, shrapnel in vital locations, surgery within 6 weeks, severe claustrophobia and severe obesity
* Previous amputation
* Life or technique expectancy < 1 year
* Pregnancy
* Peritonitis in previous 3 months
* Currently using more than one extraneal bag per 24-hours
* Known icodextrin allergy
* Currently using non-Baxter PD solutions
* Inability to provide consent
* Allergy to cholecalciferol
* Serum Calcium > 2.55 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass measured by cardiac MRI | 1 year

SECONDARY OUTCOMES:
Combined outcome of death, non-fatal CV event (stroke, MI, amputation, CHF), and transfer to HD for inadequacy or ultrafiltration failure | 3 years
Volume measures: bio-impedance (RXc graph, vector length, impedance ratio, phase angle, ECW:TBW ratio), weight, N-BNP, mean and pulse arterial pressure, number of anti-hypertensive agents | 3 years
Health-related quality of life (HRQOL) | 1 year
Physical function as measured by 6 minute walk test | 1 year
Serum and peritoneal inflammatory and fibrotic markers: albumin, CRP, IL-6, TNF-a | 1 year
Peritoneal membrane transport properties,measured by PET | 3 years
Renal and peritoneal solute clearance, 24-hour urine output and ultrafiltration volume | 3 years
left ventricular end-diastolic and systolic volumes, stroke volume and ejection fraction measure by MRI | 1 year
Fraility Score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Azim S Gangji, MD MSc FRCPC, Principal Investigator — St. Joseph's Healthcare Hamilton; K S Brimble, MD MSc FRCPC, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Population Health Research Institute - McMaster University, Hamilton, Ontario

REFERENCES:
- [Derived] Brimble KS, Ganame J, Margetts P, Jain A, Perl J, Walsh M, Bosch J, Yusuf S, Beshay S, Su W, Zimmerman D, Lee SF, Gangji AS. Impact of Bioelectrical Impedance-Guided Fluid Management and Vitamin D Supplementation on Left Ventricular Mass in Patients Receiving Peritoneal Dialysis: A Randomized Controlled Trial. Am J Kidney Dis. 2022 Jun;79(6):820-831. doi: 10.1053/j.ajkd.2021.08.022. Epub 2021 Oct 14. PMID 34656640
- [Derived] Su WS, Gangji AS, Margetts PM, Bosch J, Yusuf S, Clase CM, Ganame J, Noseworthy M, Lonn E, Jain AK, McCormick B, Brimble KS. The fluid study protocol: a randomized controlled study on the effects of bioimpedance analysis and vitamin D on left ventricular mass in peritoneal dialysis patients. Perit Dial Int. 2011 Sep-Oct;31(5):529-36. doi: 10.3747/pdi.2010.00232. Epub 2011 May 31. PMID 21632446
- See also: Hamilton Centre for Kidney Research — http://www.hamiltonkidneyresearch.ca/